CLINICAL TRIAL: NCT02503878
Title: Sedline 4 Channel Electroencephalogram (EEG) Monitoring During Suppression of Unilateral Hemispheric Function (Wada Test)
Brief Title: Sedline 4 Channel Electroencephalogram (EEG) Monitoring During Suppression of Unilateral Hemispheric Function (Wada Test
Status: Terminated | Type: Observational
Why Stopped: There was to much artifact on the readings and could not be interpreted
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, William Hand, Assistant Professor, Medical University of South Carolina
Other Study IDs: Pro00037965
Record Dates: First submitted 2015-07-17; First posted 2015-07-21 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-02

CONDITIONS: Seizure
MeSH Terms: conditions — Seizures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Masimo Sedline brain function monitors — Masimo Sedline brain function monitors are sensors (stickers) placed on a the forehead to monitor levels of "sedation" based on a bilateral 4-channel electroencephalogram (EEG). The purpose of this study is to observe the effectiveness of the Sedline monitor to detect the unilateral hemispheric EEG changes seen in Wada testing

SUMMARY:
Masimo Sedline brain function monitors are sensors (stickers) placed on a the forehead to monitor levels of "sedation" based on a bilateral 4-channel electroencephalogram (EEG). The purpose of this study is to observe the effectiveness of the Sedline monitor to detect the unilateral hemispheric EEG changes seen in Wada testing

ELIGIBILITY:
Inclusion Criteria:

18 years of age or older

scheduled for Wada testing at MUSC

Exclusion Criteria:

No exclusions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be 10 adult patients over 18 years old scheduled for Wada Testing at MUSC. One of the study team members will inform patients scheduled to undergo surgery about the opportunity to participate in the study prior to surgery. Patients will review and sign a written informed consent with a research study team member.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2014-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Masimo Sedline brain function monitor- based on a bilateral 4-channel electroencephalogram (EEG). The purpose of this study is to observe the effectiveness of the Sedline monitor to detect the unilateral hemispheric EEG changes seen in Wada testing | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States